CLINICAL TRIAL: NCT02456909
Title: The Effect of Patient Controlled Analgesia Pump Cues on Patient Satisfaction
Brief Title: Patient Controlled Analgesia Pump Cues on Patient Satisfaction
Acronym: PCA Cues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Keri Hainsworth, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NICU_RCT
Record Dates: First submitted 2015-04-27; First posted 2015-05-29 (Estimated); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cues (Experimental): The PCA pump will be programmed to provide a cue to the end of the lockout period.
  Interventions: Device: Patient-Controlled Analgesia pump with Cues; Drug: Morphine
- No Cues (Placebo Comparator): The PCA pump will be programmed such that no cues will be provided to the end of the lockout period (current standard of care).
  Interventions: Device: Patient-Controlled Analgesia pump without Cues; Drug: Morphine

INTERVENTIONS:
Device: Patient-Controlled Analgesia pump with Cues — The end of the lockout period will be cued via the PCA pump
  Arms: Cues
Device: Patient-Controlled Analgesia pump without Cues — The PCA pump will be programmed such that no cues will be provided to the end of the lockout period.
  Arms: No Cues
Drug: Morphine — Morphine will be administered for post-operative pain in both the Cues and Non-Cues groups

SUMMARY:
To examine whether providing patients with a cue to the availability of pain medication affects patient satisfaction, patient anxiety, PCA efficacy, and safety.

DETAILED DESCRIPTION:
Post-operative pain is primarily managed via Patient-Controlled Analgesia (PCA). The newest PCA pumps can be programmed so that the button is backlit with a green light at the end of the lockout period, and the green light flashes when the medication is being dispensed. No studies have examined whether this type of visual cue would influence satisfaction or other patient outcomes (such as opioid consumption, PCA safety and patient anxiety) in children and adolescents, and no studies have examined whether pediatric patients' perspectives would be similar to those of adults.

ELIGIBILITY:
Inclusion Criteria:

* 7-18 years
* Opioid naïve
* Scheduled for a surgery for which a PCA is routinely used for post-operative pain management
* At least 1 parent speaks English

Exclusion Criteria:

* Prior experience with PCA
* Cognitive delay precluding independent use of the PCA button
* Current use of anxiolytics or antidepressants
* Patients receiving epidural analgesia

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2015-04; Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keri R. Hainsworth, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants could not be recruited after surgery; therefore, all eligible participants were recruited, but not all received a PCA after surgery.
Period: Overall Study
Arm/Group | Cues | No Cues
Started | 88 | 88
Completed | 64 | 61
Not Completed | 24 | 27
Not completed — Did not receive allocated intervention | 24 | 26
Not completed — Did not complete the primary outcome | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cues | No Cues | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 61 | 125
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 61 | 125
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11 [9.0 to 11.5] | 11 [9.0 to 12.0] | 11 [9.0 to 12.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 58 | 52 | 110
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 8 | 16
  White | 48 | 47 | 95
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction Questionnaire
Description: Patient satisfaction with their PCA pump. Satisfaction was measured on a 0 to 10 scale, with higher numbers indicating greater satisfaction.
Time Frame: Up to 72 hours
Population: Includes participants who completed the post-intervention survey.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cues | No Cues
Number analyzed (Participants) | 60 | 60
units on a scale | 8 [6 to 9] | 7.5 [5 to 9]

2. Secondary Outcome: Opioid Consumption (Total Amount of Opioid Consumed Post-operatively)
Description: Total amount of opioid consumed post-operatively in mg/kg/hour.
Time Frame: Post-op Days [POD] 0 - 2, up to 72 hours
Measure: Median (Inter-Quartile Range); unit: mg/kg/hr
Arm/Group | Cues | No Cues
Number analyzed (Participants) | 64 | 61
mg/kg/hr
  Post-op Day 0 | 0.0252 [0.015 to 0.038] | 0.0248 [0.015 to 0.034]
  Post-op Day 1 | 0.0214 [0.012 to 0.031] | 0.0163 [0.011 to 0.028]
  Post-op Day 2 | 0.0162 [0.0045 to 0.024] | 0.0125 [0.0057 to 0.023]

3. Secondary Outcome: Anxiety (State Anxiety on POD 1 and POD 2)
Description: State anxiety on POD 1 and POD 2. The total score is presented as a T-score, which ranges from 0 to 100, with higher scores indicating greater levels of state anxiety. With a T-score, the mean is always 50, and the standard deviation is always 10.
Time Frame: Up to 72 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cues | No Cues
Number analyzed (Participants) | 64 | 61
units on a scale
  POD 1 | 55 [48.00 to 62.00] | 55 [49.00 to 60.00]
  POD 2 | 53.5 [46.00 to 61.00] | 52 [46.00 to 58.50]

ADVERSE EVENTS:
Time Frame: 72 hours
Description: Deaths were not assessed in this protocol.
Arm/Group | Cues | No Cues
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/62
Other Adverse Events (participants affected / at risk) | 11/64 | 6/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cues (N=64) | No Cues (N=62)
Itching requiring treatment on POD 0 (Skin and subcutaneous tissue disorders) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT02456909/Prot_SAP_000.pdf